CLINICAL TRIAL: NCT00918918
Title: The Effect of Moderate Alcohol Consumption on a Human in Vivo Model of Low-grade Systemic Inflammation in Young, Normal-weight Men
Brief Title: Effect of Alcohol Consumption on Markers of Inflammation
Acronym: AR23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Henk Hendriks, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P8600
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Alcohol Consumption; Inflammation
Keywords: Alcohol Consumption; High Density Lipoprotein (HDL); lipopolysaccharides (LPS); Apolipoproteins; Inflammation
MeSH Terms: conditions — Alcohol Drinking; Inflammation | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment B (Experimental): Vodka + orange juice
  Interventions: Dietary Supplement: Alcohol + orange juice
- Treatment A (Placebo Comparator): Orange juice
  Interventions: Dietary Supplement: Orange juice

INTERVENTIONS:
Dietary Supplement: Alcohol + orange juice — 100 mL Vodka (37.5 vol%; 30 gram of alcohol/day) + 200 mL orange juice
  Arms: Treatment B
Dietary Supplement: Orange juice — 200 mL orange juice
  Arms: Treatment A

SUMMARY:
Rationale: High-density lipoprotein (HDL), which is consistently increased after moderate alcohol consumption, is an abundant plasma lipoprotein that is generally thought to be anti-inflammatory in both health and infectious disease. HDL binds and neutralizes the bioactivity of potent bacterial remnants such as lipopolysaccharides (LPS) which stimulate the host innate immune responses.

Primary objective: To explore whether prolonged moderate alcohol consumption affects in vivo cytokine response after a low dose of LPS in young, normal-weight men.

DETAILED DESCRIPTION:
Cytokine response in a human model of low-grade systemic inflammation Lipopolysaccharide (LPS) or endotoxin is a constituent of the Gram-negative bacterial cell wall. It circulates in the plasma of healthy human subjects at low concentrations (between 1 and 200 pg/mL). Furthermore, the human gut is host to ~100 trillion organisms, which together contribute to an enteric reservoir of ~1 g LPS (4).

Upon introduction in the bloodstream endotoxin binds to LPS-binding protein (LBP) and this complex binds to CD14 on monocytes. CD14 does not have an intracellular domain but signals through Toll-like receptor 4, leading eventually to activation of the transcription factor NF-κB and to production of Tumor Necrosis Factor alpha (TNF-α,) and interleukin 6 (IL-6) and a systemic inflammatory response.

Endotoxin administration to humans, when given in a low dose, is a well-established model of systemic inflammation (5). The low dose of endotoxin elicits an acute mild systemic inflammation with a significant and reproducible cytokine and leucocyte response without increases in body temperature (2;3). This model thus resembles the levels reported in chronic low-grade inflammatory conditions such as type 2 diabetes and arthrosclerosis.

High-density lipoprotein (HDL) is a group of lipoprotein particles which have the highest density in the circulation. HDL has several anti-atherogenic effects, including the ability to transport excess cellular cholesterol to the liver for excretion, to protect low-density lipoprotein (LDL) against oxidation and to inhibit platelet aggregation. Besides its pivotal role in protecting against atherosclerosis, accumulating evidence also suggest that HDL possesses anti-inflammatory effects and plays an important role in modulating the inflammatory response to lipopolysaccharides.

Although all lipoprotein classes have been demonstrated to bind LPS, when added to whole human normal blood, it mainly binds to HDL (60%), in addition to LDL (25%) and VLDL (12%) (6). In vitro, LPS bound to lipoprotein was 20- to 1000-fold less active than the unbound form in inducing monocytes and macrophages to release cytokines (7). When transgenic mice with 2-fold elevation of plasma HDL levels were injected with LPS, they had more LPS bound to HDL, lower plasma cytokine levels, and improved survival rates compared with control mice (8). In humans Ex vivo reconstituted HDL abolished the LPS-induced overproduction of cytokines in patients with severe cirrhosis and controls (9) and intravenous infusion of reconstituted HDL protected humans from the toxic effects of LPS (10).

It has never been studied whether the alcohol-induced increase in HDL could attenuate the effects of LPS on cytokine response both ex vivo and in vivo. Given the fact that alcohol induces an increase in HDL (1) and that HDL has LPS-neutralizing properties, it is hypothesized that moderate alcohol consumption attenuates the LPS-induced cytokine response of TNF-α and IL-6 in young, normal-weight men.

In addition, because HDL causes down regulation of CD14 expression in monocytes (10) and because CD14 modulates the pro-inflammatory response to LPS (11), the effects of HDL on CD14 expression and expression of other genes related to inflammation will be determined in monocytes over time after both in vivo and ex vivo LPS administration. Since HDL also affects endothelial function (12;13) and since eicosanoids are important messengers during systemic inflammatory processes (14) these markers will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the health and lifestyle questionnaire (P8600 F02), physical examination and results of the pre-study laboratory tests
2. Males aged 21-40 years at Day 01 of the study.
3. Body Mass Index (BMI) of 18 - 27 kg/m2.
4. Alcohol consumption ≥ 5 and ≤ 28 standard units/week.
5. Normal eating habits as assessed by P8600 F02.
6. Voluntary participation.
7. Having given written informed consent.
8. Willing to comply with the study procedures, including refrain from drinking alcoholic drinks other then the alcoholic beverage provided by TNO during the entire study and refrain from fermented dairy and probiotics-containing products.
9. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years.
10. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from participation:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study.
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances.
3. Having a history of medical or surgical events or disease that may significantly affect the study outcome, particularly metabolic or endocrine disease and gastrointestinal disorders.
4. Use of medication that may affect the outcome of the study parameters.
5. Having a family history of alcoholism.
6. Smoking.
7. Not having appropriate veins for blood sampling/cannula insertion according to TNO.
8. Reported unexplained weight loss or gain in the month prior to the pre-study screening.
9. Reported slimming or medically prescribed diet.
10. Reported vegan, vegetarian or macrobiotic.
11. Recent blood donation (<1 month prior to the start of the study).
12. Not willing to give up blood donation during the study.
13. Personnel of TNO Quality of Life, their partner and their first and second degree relatives.
14. Not having a general practitioner.
15. Not willing to accept information transfer which concerns participation in the study, or information regarding health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.
16. Not willing your general practitioner to be notified upon participation in this study

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
In vivo cytokine response after low-dose LPS challenge | December 2009

SECONDARY OUTCOMES:
de novo adiponectin protein synthesis | December 2010
changes in microbiota | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Netherlands

REFERENCES:
- [Derived] Joosten MM, Schrieks IC, Hendriks HF. Effect of moderate alcohol consumption on fetuin-A levels in men and women: post-hoc analyses of three open-label randomized crossover trials. Diabetol Metab Syndr. 2014 Feb 18;6(1):24. doi: 10.1186/1758-5996-6-24. PMID 24548643